CLINICAL TRIAL: NCT04317235
Title: Ropivacaine for Ultrasound-guided Interscalene Block: 3mL Provide Similar Analgesia to 5mL With Less Diaphragmatic Paralysis in Shoulder Arthroscopy Surgeries
Brief Title: Ultrasound-guided Interscalene Block:3mL Ropi Provide Similar Analgesia to 5mL and Less Diaphragmatic Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint George Hospital (Other)
Responsible Party: Principal Investigator, Hazem Kafrouni, Assistant professor, Saint George Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SaintgeorgeH
Record Dates: First submitted 2019-01-23; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Diaphragmatic Paralysis
MeSH Terms: conditions — Respiratory Paralysis | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 ml ropivacaine (Active Comparator): interscalene block using 3 ml under ultrasound put medication on each nerve
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- 5 ml ropivacaine (Active Comparator): interscalene block using 5 ml under ultrasound put medication on each nerve
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — Is to put 3 ml or 5 ml and show the difference
  Other Names: interscalene

SUMMARY:
Ropivacaine for ultrasound-guided interscalene block: 3mL provide similar analgesia to 5mL with less diaphragmatic paralysis in shoulder arthroscopy surgeries

DETAILED DESCRIPTION:
Ropivacaine for ultrasound-guided interscalene block: 3mL provide similar analgesia to 5mL with less diaphragmatic paralysis in shoulder arthroscopy surgeries with no toxicity and no adverse reaction or complications we targeted under echography each nerve to be blocked alone either to put around all the nerves a big volume

ELIGIBILITY:
Inclusion Criteria:

* ASA1-2

Exclusion Criteria:

* ASA3-4 anticoagulant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic paralysis | Up to 48 hours
  on x ray we look if there is an elevated diaphragm
Pain relief | up to day 2 after operation
  pain scale 1-10 score 1 no pain and 10 severe pain first by visiting patient before discharge twice and thereafter on the phone

CONTACTS AND LOCATIONS:
Overall Officials: hazem kafrouni, Principal Investigator — Saint George Hospital

IPD SHARING:
Plan to Share IPD: No